CLINICAL TRIAL: NCT04845399
Title: A Single-Arm, Multicenter, Open-label Phase III Expansion Trial Evaluating Safety and Efficacy of Recombinant Human Coagulation Factor VIII-Fc Fusion Protein for Injection (FRSW107) in Adolescent and Adult Patients With Hemophilia A
Brief Title: Phase III Expansion Trial for Determining the Safety and Efficacy of Recombinant Human Coagulation Factor VIII-Fc Fusion Protein for Injection in Adolescent and Adult Patients With Hemophilia A
Acronym: RH-107-III02
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zhengzhou Gensciences Inc (Industry)
Collaborators: Jiangsu Gensciences lnc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTR20210593
Record Dates: First submitted 2021-04-09; First posted 2021-04-15 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2021-04

CONDITIONS: Hemophilia A
Keywords: Hemophilia A; Factor VIII-Fc Fusion Protein; Phase III Expansion Trial; Efficacy and Safety
MeSH Terms: conditions — Hemophilia A | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Participants will receive prophylaxis treatment with Recombinant Human Coagulation Factor VIII-Fc fusion for 6 months.
  Interventions: Drug: Recombinant Human Coagulation Factor VIII-Fc Fusion Protein for Injection

INTERVENTIONS:
Drug: Recombinant Human Coagulation Factor VIII-Fc Fusion Protein for Injection — Participants received prophylaxis treatment at 50 IU/ kg every three days.30-50 IU/kg is recommended to administration while bleeding occurs during the experiment.

SUMMARY:
The primary objectives of the study are to further evaluate the efficacy and safety of Recombinant Human Coagulation Factor VIII-Fc Fusion Protein for Injection (FRSW107) in adolescent and adult patients with hemophilia A.

ELIGIBILITY:
Inclusion Criteria:

* Patients Who have Completed trial of RH-107-001 (previously treated patients) Previously received Recombinant Human Coagulation Factor VIII-Fc prophylactic.
* The patient and/or guardian or his or her legal representative must be able to read, understand, and provide signed informed consent, And voluntarily signed the Informed Consent Form.
* The compliance of patients appeared quite well.
* Patient who is considered by the investigators suitable for ongoing to accept previously treated.

Exclusion Criteria:

* Subjects who have not completed trial of RH-107-001or who have completed the Phase III clinical trial but not willing to continue receiving treatment.
* Subjects who did not participate in the Phase III clinical trial of RH-107-001.

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2021-06-26 (Actual); Study Completion 2021-06-26 (Actual)

PRIMARY OUTCOMES:
Annualized Bleeding Rates (ABR). | For the duration of study participation, 6 months.
  Annualized bleeding rate = (number of bleeding episodes during the efficacy, period/total number of days during the efficacy period)*365.25. The efficacy period begins with the first prophylactic dose of FRSW107 and ends with the last dose (for prophylaxis or a bleed). Surgery/rehabilitation periods are not included in the efficacy period. A bleeding episode started from the first sign of a bleed and ended no more than 72 hours after the last treatment for the bleed, within which any symptoms of bleeding at the same location or injections less than or equal to 72 hours apart were considered the same bleeding episode. Any injection to treat the bleeding episode taken more than 72 hours after the preceding one was considered the first injection to treat a new bleeding episode at the same location. Any bleeding at a different location was considered a separate bleeding episode, regardless of time from last injection.
Number of target joints. | For the duration of study participation, 6 months.
  Describe the number and percentage of cases with target joints ≥1 and their 95% confidence intervals before and after drug administration, and compare the change in the number of target joints from baseline after treatment.
Annualized Joint Bleeding Rate (AJBR) | For the duration of study participation, 6 months.
  Annualized joint bleeding rate(AJBR)can be calculated using the following formula: Number of joint bleeding episodesevents during efficacy evaluation period/(number of days in treatment period/365.25).

SECONDARY OUTCOMES:
Total Dose Required for Resolution of a Bleeding Episode. | For the duration of study participation, 6 months.
  The total dose required to resolve a bleeding episode per participant, based on the efficacy period. The efficacy period begins with the first dose and ends with the last dose (for a bleed). For 'Per bleeding episode' values, for each bleeding episode, the total dose is the sum of the doses (IU/kg) administered across all injections given to treat that bleeding episode. For 'Per participant' values, the total dose (IU/kg) used to resolve each bleed is averaged across all bleeding episodes per participant.
Number of injections required to resolve a bleeding episode. | For the duration of study participation, 6 months.
  The number of injections required to resolve a bleeding episode per participant, based on the efficacy period. The efficacy period begins with the first dose and ends with the last dose (for a bleed). All injections given from the initial sign of a bleed, until the last date/time within the bleed window are counted. The resolution of a bleed is defined as no sign of bleeding following injection for the bleed. For 'Per participant' values, the number of injections required to resolve each bleed is averaged across all bleeding episodes per participant.
Quality of life assessment. | For the duration of study participation, 6 months.
  Quality of life assessment by Haemophilia Joint Health Score(HJHS 2.1).
Score of bleeding symptoms and Vital signs. | For the duration of study participation, 6 months.
  Response to treatment with rFVIIIFc for bleeding episodes, using the 4-point bleeding response scale.
Number of participants with inhibitor development | For the duration of study participation, 6 months.
  Number of participants who developed a positive FVIII inhibitor level (≥0.6 Bethesda unit [BU]) during the study was summarized and classified as participants developing low titer inhibitor (i.e. ≤ 5.0 BU) and participants developing high titer inhibitor (i.e. > 5.0 BU).
Number of Participants With Incidence of Antibody Formation to CHINESE HAMSTER OVARY (CHO). | For the duration of study participation, 6 months.
  A test to analyze the formation of antibodies to CHO.
Number of Participants With Adverse Events (AEs) and Serious Adverse Events. (SAEs) as a Measure of Safety and Tolerability. | For the duration of study participation, 6 months.
  An AE is any untoward medical occurrence that does not necessarily have a causal relationship with this treatment. An SAE is any untoward medical occurrence that at any dose: results in death; in the view of the Investigator, places the participant at immediate risk of death (a life-threatening event); requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; results in a congenital anomaly/birth defect; any other medically important event that, in the opinion of the Investigator, may jeopardize the participant or may require intervention to prevent one of the other outcomes listed in the definition.

CONTACTS AND LOCATIONS:
Overall Officials: Renchi Yang, Principal Investigator — Institute of Hematology & Blood Diseases Hospital Chinese Academy of Medical Sciences & Peking Union Medical College.
Locations (16):
- China (16):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Capital Medical University affiliated Beijing Children's Hospital, Beijing, Beijing Municipality
  - Chongqing Three Gorges Central Hospital, Chongqing, Chongqing Municipality
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangzhou
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangzhou
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Henan provincial People's Hospital, Zhengzhou, He'nan
  - Henan Cancer Hospital, Zhengzhou, He'nan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - The Affiliated Hospital of Xuzhou Medical College, Xuzhou, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - Jinan central hospital, Ji'nan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - The Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Institute of Hematology & Blood Diseases Hospital Chinese Academy of Medical Sciences & Peking Union Medical College., Tianjin, Tianjin Municipality